CLINICAL TRIAL: NCT03027453
Title: Berlin - Specific Acute Treatment in Ischemic or Haemorrhagic Stroke With Long Term Follow-up
Acronym: B-SPATIAL
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Berliner Feuerwehr (Unknown); Bundeswehrkrankenhaus Berlin (Other); DRK-Kliniken Berlin Köpenick (Unknown); Evangelisches Krankenhaus Königin Elisabeth Herzberge (Unknown); Helios Klinikum Berlin-Buch (Other); Jüdisches Krankenhaus Berlin (Unknown); Park-Klinik Weissensee (Unknown); Schlosspark-Klinik (Unknown); Unfallkrankenhaus Berlin (Other); Vivantes Auguste-Viktoria-Klinikum (Unknown); Vivantes Klinikum im Friedrichshain (Unknown); Vivantes Humboldt-Klinikum (Unknown); Vivantes Clinic Neukölln (Other); Vivantes Klinikum Spandau (Unknown)
Responsible Party: Principal Investigator, Heinrich J Audebert, Prof. Dr. med., Charite University, Berlin, Germany
Other Study IDs: B-SPATIAL
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The B-SPATIAL-Registry will provide a tool of quality assessment for stroke specific Treatments such as endovascular treatment. It will also enable the participating hospitals to compare the quality of care of their facility. At the same time, B-SPATIAL will provide an opportunity of scientific evaluation of new therapeutic procedures or specific treatments in stroke (i.e. reversal of oral anticoagulation in intracerebral hemorrhage or intravenous thrombolysis), not sufficiently investigated so far. Finally, the B-SPATIAL Registry will allow for an identification of key quality indicators that assure valid quality assessment aiming at a reduced documentation load for future quality management.

DETAILED DESCRIPTION:
1. Background

   Quality assessment of acute stroke care is organized in regional stroke registries in Germany - for the federal state of Berlin in the Berlin Stroke Registry (BSR). The current documentation of the Berlin Stroke Registry is focused on the documentation of process quality in participating hospitals.

   So far, outcome quality is only assessed by surrogate parameters such as complications and mortality during in-hospital stay. However, according to consensus recommendations, disability-free survival versus death and dependency is the most important outcome measure after acute stroke. Because of the high variability of the clinical course after stroke, this outcome is generally assessed after three months by using the modified Rankin Scale (mRS).
2. Motivation

   In early 2015, several published trials showed that mechanical thrombectomy improves the prognosis of ischemic stroke patients with acute large artery occlusion of proximal brain supplying arteries. Currently, this invasive catheter based treatment is not available in many hospitals with acute Stroke Unit. It is likely that the quality of technical procedures depends on the expertise and experience of treating interventionalists. Current studies suggest a close relationship between effectiveness of the approach and time to treatment, similar to intravenous thrombolysis. This time dependency makes prehospital triage more challenging because selection of the appropriate facility is likely to influence patient outcome.

   Intracerebral hemorrhage (ICH) is less frequent than ischemic stroke but is associated with worse prognosis. Recent studies suggest that blood pressure lowering may improve prognosis if started during the hyperacute phase of ICH. With limited scientific evidence, many patients undergo neurosurgical intervention. It remains unclear whether delivery of hemorrhagic stroke patients to hospitals with neurosurgery leads to better outcome.

   Hence, pre-hospital care with delivery to more or less specialized clinical facilities may have a crucial impact for both subtypes of stroke. The introduction of specialized stroke ambulances (Stroke Emergency Mobiles, STEMOs) opens new avenues for pre-hospital stroke diagnosis, treatment and patient triage. The effects of STEMO care are planned to be assessed by the parallel B-PROUD-Study (NCT02869386).
3. Purpose

   The B-SPATIAL-Registry will provide a tool of quality assessment for new specific treatments. It will also enable the participating hospitals to compare the quality of care of their own facility.

   Because this registry represents an quality monitoring initiative, the telephone follow-up is collected with an opt-out solution, allowing to decline participation after the patients are informed on the follow-up telephone call at discharge and through a letter send one month prior to the actual call. As written informed consent is not required, this method will facilitate a high follow-up rate particularly in patients with severe neurological deficits or treated in non-academic hospitals.

   In B-SPATIAL we want to identify key quality indicators that assure valid quality assessment despite reduced documentation load in future quality management.

   Specific Aims of the registry:
   * Assessment of proportions of patients receiving specific treatments (based on total number of eligible)
   * Evaluation of treatment specific indicators for process quality including pre-hospital care
   * Evaluation of outcome quality (survival, level of disability and quality of life after 3 months)

   Pre-specified analyses:

   Ischemic stroke
   * Intravenous hospital based tPA rate in treatment candidates
   * Time to treatment in intravenous tPA
   * Rate of secondary interhospital referral
   * Proportions of patients receiving endovascular thrombectomy
   * Time to groin puncture and reperfusion in patients with endovascular thrombectomy
   * Proportions of used devices
   * Proportions of patients with general/non general anesthesia (conscious sedation)
   * Secondary intracranial hemorrhage
   * Functional outcome according to mRS at 3 months

   Hemorrhagic stroke
   * Time to start of intravenous antihypertensive treatment
   * Time to start of PCC in patients with OAC or specific reversal of NOACs
   * Rate of surgical treatments
   * Rate of secondary interhospital referral
   * Enlargement and final volume of ICH
   * Functional outcome according to mRS at 3 months

   Data sources

   The documentation will include pre-hospital, in-hospital and post-discharge processes such as:
   * Emergency medical service (EMS)
   * Acute in-hospital stay
   * Follow-up (first choice: telephone, second choice: written questionnaire, third choice: FU regarding vital status from registration offices)
4. Patients

   In order to ensure valid analysis of treatment rates in participating hospitals, patients will be included according to the following inclusion criteria:
   * Patients with hospital main discharge diagnoses according to ICD 10: Ischemic stroke (I63) or TIA (G45.0-G45.3 and G45.5-G45.9, respectively) and

     * Onset of symptoms within 6 hours of hospital arrival
     * In patients with TIA diagnosis: Persistent neurological symptoms at hospital arrival (emergency department documentation)
   * Patients with main discharge diagnosis of intracranial hemorrhage and hospital admission within 6 hours of stroke onset.
   * Patients with other main discharge diagnoses and documented intravenous thrombolysis (OPS 8-020.8) in order to monitor the treatment rate of stroke mimics
5. Data documentation

   * Data will be entered in all participating hospitals via remote access to the databank
   * Data will be entered with pseudonyms but identification will only be possible in local hospitals via register-logs that will be safely stored in the hospitals.
6. Databank characteristics

   * For data entry, we will use the REDcap databank software with access from all participating hospitals.
   * Dedicated computers will be used and safely stored in participating hospitals. Encryption and password algorithms will protect the remote access to the databank.
   * The registry databank will be stored and hosted on a protected server of the Charité IT department.
   * For statistical evaluation, the REDcap databank will be exported in an SPSS-based data format, stored on the server of the Center for Stroke Research Berlin (CSB).
7. Responsibilities

   * Data entry: Study nurses in participating hospitals
   * Databank in Charité IT-center: Charité IT department and databank manager of the Clinical Research Units
   * Scientific evaluation: PI of CSB (Jessica L.Rohmann in cooperation with Heinrich J. Audebert, Martin Ebinger and Christian Nolte)

ELIGIBILITY:
Inclusion criteria:

1. Patients with hospital main discharge diagnoses according to ICD 10: Ischemic stroke (I63) or TIA (G45.0-G45.3 and G45.5-G45.9, respectively) and

   * Onset of symptoms within 6 hours of hospital arrival
   * In patients with TIA diagnosis: Persistent neurological symptoms at hospital arrival (emergency department documentation)
2. Patients with main discharge diagnosis of intracranial hemorrhage and symptom onset within 6 hours of hospital admission
3. Patients with other main discharge diagnoses and documented intravenous thrombolysis (OPS 8-020.8) in order to monitor the treatment rate of stroke mimics

Exclusion Critera:

* Symptom remission before EMS arrival or hospital arrival (if no EMS Transport)
* Primary subarachnoid hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients (ischemic and haemorrhagic)
Sampling Method: Non-Probability Sample
Enrollment: 15246 (Actual)
Dates: Start 2016-01; Primary Completion 2021-04 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale | 3 months
  Assessment of functional outcome over the entire range of the modified Rankin Scale

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Rohmann, Principal Investigator — Center for Stroke Research Berlin
Locations (1):
- Center for Stroke Research Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ebinger M, Winter B, Wendt M, Weber JE, Waldschmidt C, Rozanski M, Kunz A, Koch P, Kellner PA, Gierhake D, Villringer K, Fiebach JB, Grittner U, Hartmann A, Mackert BM, Endres M, Audebert HJ; STEMO Consortium. Effect of the use of ambulance-based thrombolysis on time to thrombolysis in acute ischemic stroke: a randomized clinical trial. JAMA. 2014 Apr 23-30;311(16):1622-31. doi: 10.1001/jama.2014.2850. PMID 24756512
- [Background] Krebes S, Ebinger M, Baumann AM, Kellner PA, Rozanski M, Doepp F, Sobesky J, Gensecke T, Leidel BA, Malzahn U, Wellwood I, Heuschmann PU, Audebert HJ. Development and validation of a dispatcher identification algorithm for stroke emergencies. Stroke. 2012 Mar;43(3):776-81. doi: 10.1161/STROKEAHA.111.634980. Epub 2012 Jan 5. PMID 22223240
- [Background] Ebinger M, Fiebach JB, Audebert HJ. Mobile computed tomography: prehospital diagnosis and treatment of stroke. Curr Opin Neurol. 2015 Feb;28(1):4-9. doi: 10.1097/WCO.0000000000000165. PMID 25490196
- [Background] Wendt M, Ebinger M, Kunz A, Rozanski M, Waldschmidt C, Weber JE, Winter B, Koch PM, Freitag E, Reich J, Schremmer D, Audebert HJ; STEMO Consortium. Improved prehospital triage of patients with stroke in a specialized stroke ambulance: results of the pre-hospital acute neurological therapy and optimization of medical care in stroke study. Stroke. 2015 Mar;46(3):740-5. doi: 10.1161/STROKEAHA.114.008159. Epub 2015 Jan 29. PMID 25634000
- [Background] Kunz A, Ebinger M, Geisler F, Rozanski M, Waldschmidt C, Weber JE, Wendt M, Winter B, Zieschang K, Fiebach JB, Villringer K, Erdur H, Scheitz JF, Tutuncu S, Bollweg K, Grittner U, Kaczmarek S, Endres M, Nolte CH, Audebert HJ. Functional outcomes of pre-hospital thrombolysis in a mobile stroke treatment unit compared with conventional care: an observational registry study. Lancet Neurol. 2016 Sep;15(10):1035-43. doi: 10.1016/S1474-4422(16)30129-6. Epub 2016 Jul 16. PMID 27430529
- [Derived] Rohmann JL, Huerta-Gutierrez R, Audebert HJ, Kurth T, Piccininni M. Adjusted horizontal stacked bar graphs ("Grotta bars") for consistent presentation of observational stroke study results. Eur Stroke J. 2023 Mar;8(1):370-379. doi: 10.1177/23969873221149464. Epub 2023 Jan 13. PMID 37021164